CLINICAL TRIAL: NCT00893646
Title: Effects of Weight Reduction and Lifestyle Changes on Sleep, Alertness and Cardiometabolic Risk Factors in Overweight Professional Long-distance Drivers
Brief Title: Effects of Weight Reduction on Sleep and Alertness in Long-distance Truck and Bus Drivers
Acronym: SF-Truck
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UKK Institute (Other)
Collaborators: Academy of Finland (Other); Finnish Institute of Occupational Health (Other); Vitalmed Research Centre (Other)
Responsible Party: Principal Investigator, Katriina Kukkonen-Harjula, senior researcher, UKK Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R09025; SA124344
Record Dates: First submitted 2009-05-04; First posted 2009-05-06 (Estimated); Last update posted 2015-06-01 (Estimated); Status verified 2015-05

CONDITIONS: Abdominal Obesity
Keywords: abdominal obesity; weight reduction; diet; exercise training; lifestyle activity; health-related fitness; walking; actigraphy; lifestyle modification; sleep; sleep hygiene; alertness; daytime sleepiness; metabolic syndrome; counselling; health education; truck drivers; bus drivers; randomized controlled trial
MeSH Terms: conditions — Obesity, Abdominal; Weight Loss; Sleep Hygiene; Disorders of Excessive Somnolence; Metabolic Syndrome; Health Education

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- weight loss counseling (Experimental): individual monthly counseling on diet, physical activity and sleep
  Interventions: Behavioral: weight loss counseling
- control (No Intervention): no lifestyle advice, yearly assessments

INTERVENTIONS:
Behavioral: weight loss counseling — individual monthly lifestyle counseling, face-to-face (6 times, each 45 min) and by telephone (7 times, each 30 min), on how to decrease energy intake and change eating habits to improve quality of dietary fat and carbohydrate, how to increase daily walking steps; and how to improve sleep quality (sleep hygienic tips)
  Other Names: lifestyle counseling
  Arms: weight loss counseling

SUMMARY:
The study is a year-long health-behaviour intervention in obese, male truck-drivers to lose weight moderately by 10%, using monthly individual counseling. The investigators hypothesize that lifestyle modification (increased physical activity, changes in eating habits, and improved schedule for sleep) through weight loss improves daytime alertness and quality of sleep, reduces daytime sleepiness, and improves cardiovascular risk factors and health-related fitness.

DETAILED DESCRIPTION:
Daytime sleepiness, i.e., being fatigued at work is an important risk factor for traffic accidents involving commercial vehicles. Sleep-related disturbances and daytime fatigue may be partly related to obesity, which is common among truck drivers. This study is a randomised 12-month health-behaviour intervention in obese, male truck-drivers. We hypothesize that lifestyle modification (increased physical activity; decreased energy intake; and improved schedule for sleep), aimed to reduce weight moderately by 10%, improves daytime alertness and quality of sleep, reduces daytime sleepiness, and improves cardiometabolic health and health-related fitness. The primary aim is weight loss. We will recruit 140 participants aged 30-62 years and with abdominal obesity. The participants are randomised into an intervention (INT) and control (CON) group, for 12 months. The INT group gets individual lifestyle counseling monthly. After 12 months, the CON group receives weight-loss counseling for 3 months. Assessments (psychological vigilance test, sleep duration, dietary intake, physical activity, metabolic syndrome, health-related fitness) take place at months 0, 12 and 24. We expect to develop counseling strategies (leading to weight loss through changes in lifestyle) that can be used to improve sleep, alertness and cardiometabolic health in occupational health care.

ELIGIBILITY:
Inclusion Criteria:

* male
* age 30-62 years
* long-distance truck or bus driver (on average continuous driving for at least one hour daily outside the city center)
* irregular working hours (on average at least once weekly between 0600-1800 hours)
* waist circumference at least 100 cm
* sedentary: leisure physical activity no more than 30 minutes twice weekly at moderate intensity, and no medical contraindications to increase physical activity

Exclusion Criteria:

* no moderate or severe sleep apnoea with CPAP therapy or with previous surgical operations in the neck area (e.g., UPPP)
* no regular use of sleeping medicines (on average not more often than once weekly)
* no severe sleep disorder
* greatly elevated resting blood pressure (> 180/120 mmHg)
* no diabetes mellitus with medication

Ages: 30 Years to 62 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 113 (Actual)
Dates: Start 2009-05; Primary Completion 2012-06 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
body weight | 12 months

SECONDARY OUTCOMES:
sleep duration | 12 months
alertness (ability to stay awake) | 12 months
occurrence of metabolic syndrome | 12 months
health-related fitness | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Katriina T Kukkonen-Harjula, MD, Ph.D., Principal Investigator — UKK Institute for Health Promotion Research
Locations (3):
- Finland (3):
  - Finnish Institute of Occupational Health, Helsinki
  - Vitalmed Research Centre & Sleep Clinic, Helsinki
  - UKK Institute for Health Promotion Research, Tampere

REFERENCES:
- [Derived] Puhkala J, Kukkonen-Harjula K, Aittasalo M, Mansikkamaki K, Partinen M, Hublin C, Karmeniemi P, Sallinen M, Olkkonen S, Tokola K, Ojala A, Nygard CH, Fogelholm M. Lifestyle counseling in overweight truck and bus drivers - Effects on dietary patterns and physical activity. Prev Med Rep. 2016 Aug 15;4:435-40. doi: 10.1016/j.pmedr.2016.08.012. eCollection 2016 Dec. PMID 27583202